CLINICAL TRIAL: NCT06792474
Title: Influence of Lidocaine Infusion on Motor Evoked Potential Thresholds; a Single-center, Double-blinded, Randomized Trial for Patients Undergoing Spin Surgery With Intraoperative Neurophysiologic Monitoring.
Brief Title: Influence of Lidocaine Infusion on Motor Evoked Potential Thresholds
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Lauren K. Buhl, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY02002708
Record Dates: First submitted 2024-12-26; First posted 2025-01-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Spinal Disease; Anesthesia; Post Operative Pain
Keywords: Lidocaine; Intraoperative Neuromonitoring; Spine surgery; Post Operative Pain
MeSH Terms: conditions — Spinal Diseases; Pain, Postoperative | interventions — Lidocaine; Sodium Chloride; Exercise; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single-center, double-blinded, randomized trial with randomization to lidocaine infusion or saline infusion for patients undergoing spine surgery with intraoperative neurophysiological monitoring
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Research Pharmacy will compound lidocaine 2,000 mg (4 mg/mL) in 500 mL 0.9% sodium chloride or placebo (infusion bags will be aseptically prepared in a biological safety cabinet.) The lidocaine or placebo bags will be delivered and stored in the Same Day Procedure Omnicell machine prior to the day of procedure. The infusion bags will not be labeled as lidocaine or placebo in order not to unblind the blinded personnel administering the investigational product and will contain the calculated rate of infusion.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine Infusion (Active) (Active Comparator): Lidocaine infusion
  Interventions: Drug: Lidocaine in Saline
- Normal Saline Infusion (Sham) (Sham Comparator): Normal saline infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine in Saline — Lidocaine infusion 1.5 mg/kg/hr
  Other Names: Active
  Arms: Lidocaine Infusion (Active)
Drug: Normal saline — Normal saline infusion
  Other Names: Placebo
  Arms: Normal Saline Infusion (Sham)

SUMMARY:
The purpose of this study is to determine the effect of lidocaine infusion on intraoperative neuromonitoring in patients undergoing spine surgery.

DETAILED DESCRIPTION:
The investigators will compare the stimulation threshold for motor evoked potentials (MEPs) for patients undergoing spine surgery with intraoperative neurophysiologic monitoring (IONM) who receive a lidocaine infusion vs. normal saline (NS) infusion. The endpoint for this objective will be the final stimulation threshold for MEPs at the end of the surgery. The stimulation threshold for MEPs is a commonly used metric to determine the effects of anesthetic agents on MEP signals. Secondary objectives will somatosensory evoked potentials (SSEPs) with an endpoint of amplitude and latency of SSEPs throughout the surgery. Other secondary outcomes will include, intraoperative mean arterial pressure (MAP), intraoperative propofol consumptions, and post-operative visual analog scale (VAS) and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cervical or thoracolumbar spine surgery with intraoperative neurophysiological monitoring

Exclusion Criteria:

* Inability to provide informed consent in English
* Pregnancy (based on patient report or a positive test on the day of surgery)
* Contraindication to lidocaine
* Planned post-operative intubation
* Current incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potentials (MEPs) | Duration of the surgical procedure, no more than 24 hours
  An endpoint of the final stimulation threshold for MEPs at the end of surgery.

SECONDARY OUTCOMES:
Somatosensory Evoked Potentials (SSEPs) | Duration of the surgical procedure, no more than 24 hours
  Endpoints of amplitude and latency throughout the surgery of SSEPs
Mean Arterial Pressure (MAP) | Duration of the surgical procedure, no more than 24 hours
  Intraoperative incidence of MAP <65 mmHg and MAP < 55 mmHg
Intraoperative propofol consumption | Duration of the surgical procedure, no more than 24 hours
  Rate of propofol consumption between the arms
Visual Analog Scale (VAS) Pain Scores | Post-operative day 0 through 3
  Endpoint of VAS pain scores post operative days (POD) 0/1/3
Opiod consumption | Post-operative day 0 through 3
  Opiod consumption converted to morphine equivalents through post operative day (POD) 3

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sloan TB, Mongan P, Lyda C, Koht A. Lidocaine infusion adjunct to total intravenous anesthesia reduces the total dose of propofol during intraoperative neurophysiological monitoring. J Clin Monit Comput. 2014 Apr;28(2):139-47. doi: 10.1007/s10877-013-9506-x. Epub 2013 Aug 31. PMID 23996498
- [Background] Urban MK, Fields K, Donegan SW, Beathe JC, Pinter DW, Boachie-Adjei O, Emerson RG. A randomized crossover study of the effects of lidocaine on motor- and sensory-evoked potentials during spinal surgery. Spine J. 2017 Dec;17(12):1889-1896. doi: 10.1016/j.spinee.2017.06.024. Epub 2017 Jun 27. PMID 28666848
- [Background] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Background] Leliefeld PH, Wessels CM, Leenen LP, Koenderman L, Pillay J. The role of neutrophils in immune dysfunction during severe inflammation. Crit Care. 2016 Mar 23;20:73. doi: 10.1186/s13054-016-1250-4. PMID 27005275
- [Background] Karnina R, Arif SK, Hatta M, Bukhari A. Molecular mechanisms of lidocaine. Ann Med Surg (Lond). 2021 Aug 17;69:102733. doi: 10.1016/j.amsu.2021.102733. eCollection 2021 Sep. PMID 34457261
- [Background] Hollmann MW, Herroeder S, Kurz KS, Hoenemann CW, Struemper D, Hahnenkamp K, Durieux ME. Time-dependent inhibition of G protein-coupled receptor signaling by local anesthetics. Anesthesiology. 2004 Apr;100(4):852-60. doi: 10.1097/00000542-200404000-00015. PMID 15087620
- [Background] Dewinter G, Moens P, Fieuws S, Vanaudenaerde B, Van de Velde M, Rex S. Systemic lidocaine fails to improve postoperative morphine consumption, postoperative recovery and quality of life in patients undergoing posterior spinal arthrodesis. A double-blind, randomized, placebo-controlled trial. Br J Anaesth. 2017 Apr 1;118(4):576-585. doi: 10.1093/bja/aex038. PMID 28403408
- [Background] Farag E, Ghobrial M, Sessler DI, Dalton JE, Liu J, Lee JH, Zaky S, Benzel E, Bingaman W, Kurz A. Effect of perioperative intravenous lidocaine administration on pain, opioid consumption, and quality of life after complex spine surgery. Anesthesiology. 2013 Oct;119(4):932-40. doi: 10.1097/ALN.0b013e318297d4a5. PMID 23681143
- [Background] Schubert A, Licina MG, Glaze GM, Paranandi L. Systemic lidocaine and human somatosensory-evoked potentials during sufentanil-isoflurane anaesthesia. Can J Anaesth. 1992 Jul;39(6):569-75. doi: 10.1007/BF03008320. PMID 1386560